CLINICAL TRIAL: NCT06814197
Title: Reducing Procrastination With One-to-One, Lay-Delivered Teletherapy: Protocol for A Mixed-Methods, Waitlist-Controlled Trial
Brief Title: Overcoming Procrastination in Adults: A Waitlist-Controlled Trial of One-to-One Online Coaching With Trained Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Overcome (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P-PF-11.24.0004
Record Dates: First submitted 2025-01-17; First posted 2025-02-07 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Procrastination
Keywords: Procrastination; Motivational Interviewing; Cognitive Behavioural Therapy; Behaviour Change; CBT; MI; Randomised Controlled Trial; RCT; Lay Counselling; Teletherapy; eHealth; Coaching
MeSH Terms: interventions — Motivational Interviewing; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Intervention Group: Participants will receive the intervention immediately.
  Waitlist Control Group: Participants will be on a four-week waitlist. They will receive the intervention after completing their participation in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motivational Interviewing and Cognitive Behavioural Therapy for Procrastination (Experimental): A 4-week intervention will be delivered remotely via Zoom or Google Meets, guided by Overcome coaches. Coaches are trained over two days via training slides, role plays and feedback. The intervention incorporates Motivational Interviewing and Cognitive Behavioural Therapy.
  Interventions: Behavioral: Motivational Interviewing and Cognitive Behavioural Therapy for Procrastination
- Waitlist Control (No Intervention): Participants will be on the waitlist for four weeks and complete outcome measures. After they have completed the outcome measures and concluded their participation in the study, they will receive the intervention too.

INTERVENTIONS:
Behavioral: Motivational Interviewing and Cognitive Behavioural Therapy for Procrastination — This intervention incorporates Motivational Interviewing (e.g., open-ended questions, affirmations, reflective listening, summarising) and Cognitive Behavioural Therapy (e.g., cognitive restructuring) techniques in natural conversations instead of having a fully manualised programme. This approach resembles coaching instead of traditional therapy to build therapeutic relationships naturally and keep clients engaged with genuine human connection.
  Arms: Motivational Interviewing and Cognitive Behavioural Therapy for Procrastination

SUMMARY:
The goals of this clinical trial are to assess the feasibility and efficacy of a one-to-one, layperson-delivered, online Motivational Interviewing (MI) and Cognitive Behavioral Therapy (CBT) intervention for adults aged 18 to 64 experiencing severe procrastination but without moderate-to-severe anxiety or depression.

The main questions it aims to answer are:

* Can a layperson-delivered, online MI and CBT intervention effectively reduce procrastination compared to a waitlist control group?
* Can the intervention effectively improve self-efficacy and life satisfaction?
* Are the effects of the intervention maintained one month after completion?

Eligible participants will be randomly assigned to either the Intervention group or the Waitlist Control group, with baseline procrastination, self-efficacy, and life satisfaction measured beforehand. Participants in the intervention group will attend four weekly 60-minute online sessions delivered by trained lay coaches supervised by experienced specialists. Sessions will focus on goal-setting, identifying triggers, improving time management, and creating long-term plans to sustain progress. At the end of the intervention, 12 participants will be interviewed to share their experiences. Participants in the waitlist control group will continue their usual activities for four weeks and will receive the same intervention after completing the study assessments. This group will serve as a comparison to evaluate the effectiveness of the intervention.

DETAILED DESCRIPTION:
Procrastination is a prevalent behavioural issue affecting around 20% of adults, leading to decreased productivity, financial losses, and adverse mental health outcomes such as increased stress and reduced life satisfaction. Despite these significant effects, it is often overlooked in mental health services and under-researched as a condition requiring targeted interventions.

Cognitive Behavioural Therapy (CBT) has been the primary approach used to address procrastination, focusing on restructuring maladaptive beliefs, goal setting, and increasing task engagement. However, most existing studies focus on therapist-led interventions, making these treatments costly and less scalable. Motivational Interviewing (MI) complements CBT by addressing low self-efficacy and enhancing commitment to behavioural change through client-centred techniques such as reflective listening and eliciting "change talk". Layperson-delivered interventions, which involve non-clinicians providing structured support, have shown promise in making therapies more accessible and cost-effective.

There is limited research on scalable, lay-delivered procrastination interventions, particularly those combining CBT and MI techniques in a remote format. This study aims to address this gap by evaluating the efficacy and feasibility of a four-week online, one-to-one intervention.

The primary objectives are to:

* Measure changes in procrastination, self-efficacy, and life satisfaction.
* Assess the feasibility of delivering the intervention, focusing on recruitment, adherence, and participant satisfaction.

This is a mixed-methods, waitlist-controlled trial. Participants are randomly allocated to either an Intervention or Waitlist Control group. The intervention involves four weekly 60-minute video sessions delivered by trained lay coaches. The waitlist control group will receive the intervention after a four-week waitlist period.

Participants will be adults aged 18 to 64 with severe procrastination (Irrational Procrastination Scale [IPS] ≥ 32) but without moderate-to-severe anxiety or depression (PHQ-9 < 15 and GAD-7 < 12). Exclusion criteria include cognitive impairments, severe psychiatric diagnoses, and significant health conditions. Participants will complete an online screening questionnaire and a follow-up call to confirm eligibility. After providing informed consent, participants will be randomised using block randomisation to ensure balanced group distribution.

Quantitative data will be collected at baseline, post-intervention, and at a one-month follow-up for the intervention group. Qualitative data will be gathered through post-intervention interviews with 12 participants, using thematic analysis to explore experiences and engagement. Statistical analysis will include two-way repeated measures ANOVAs and exploratory mediation models to evaluate changes in key outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 64.
* Access to a computer or mobile device with internet connectivity.
* Ability to understand and speak English.
* IPS score ≥ 32 to confirm severe procrastination.
* PHQ-9 score < 15 to exclude moderate-to-severe depressive symptoms.
* GAD-7 score < 12 to exclude moderate-to-severe anxiety symptoms.

Exclusion Criteria:

* Cognitive impairments, significant health conditions or disabilities affecting the ability to provide consent and fully participate.
* Psychiatric diagnoses requiring specialist care (e.g., schizophrenia, eating disorders, substance misuse). Such participants will be signposted to relevant local services if needed.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Change in Irrational Procrastination Scale (IPS) | From enrolment to one-month follow-up (8 weeks in total).
  Irrational Procrastination Scale is a self-report questionnaire measuring procrastination with 9 items on a 5-point Likert scale from 1 (Very Self or Not True of Me) to 5 (Very Often True, or True of Me). The total score is obtained by adding up the scores of each response, with three items reverse-coded. The total score ranges from 9 to 45. IPS has good internal consistency, strong reliability and concurrent validity for use across diverse populations. administered at sign-up, post-intervention, and at one-month follow-up to monitor the effectiveness of the intervention.

SECONDARY OUTCOMES:
Change in General Self-Efficacy Scale (GSE) | From enrolment to one-month follow-up (8 weeks in total).
  General Self-Efficacy Scale is a self-report questionnaire measuring self-efficacy with 10 items on a 4-point Likert scale from 1 (Not at all true) to 4 (Exactly true), with the total score ranging from 10 to 40. General Self-Efficacy Scale has good internal consistency, strong reliability and concurrent validity for use across different settings and groups. General Self-Efficacy Scale is a secondary measure of this study, administered at sign-up, post-intervention, and at one-month follow-up.
Change in Cantril Ladder | From enrolment to one-month follow-up (8 weeks in total).
  Cantril Ladder measures life satisfaction on an 11-point Likert scale from 0 (Worst possible life) to 10 (Best possible life). Cantril Ladder has good internal consistency, strong reliability and concurrent validity for use across different populations. Cantril Ladder is a secondary measure of this study, administered at sign-up, post-intervention, and at one-month follow-up.

OTHER OUTCOMES:
Enrollment rate | From the screening call to the time of enrolment in the study, with follow-up for up to 2 weeks after the screening call.
  The number of participants who enrolled in the study (i.e., signed the consent form) after attending the screening call, out of the total number of participants deemed eligible to participate in the study (based on inclusion and exclusion criteria) after the screening call. A higher percentage indicates a more effective enrolment process.
Eligibility rate | From the screening call to when eligibility is confirmed, within 2 days after the screening call.
  The number of participants deemed eligible to participate in the study (based on inclusion and exclusion criteria) after the screening call, out of the total number of participants who attended the screening call. A higher percentage reflects a more targeted recruitment strategy.
Attrition | From enrolment to post-intervention interview (5 weeks in total).
  Number of individuals who dropped out (dropouts only). The study aims to achieve lower attrition rates.
Adherence | From enrolment to last session (4 weeks in total).
  Number of intervention sessions attended. The higher number is the desired outcome.
Satisfaction with the intervention | Post-intervention interview (Week 5).
  Participants will rate their satisfaction with the remotely delivered intervention (10-point Likert scale from 1 to 10). The higher ratings are more desirable outcomes.
Perceived engagement with the intervention | Post-intervention interview (Week 5).
  Participants will rate their perceived engagement with the remotely delivered intervention (10-point Likert scale from 1 to 10). The higher ratings are more desirable outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Overcome, Arnside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The researchers decided not to make the IPDs shareable to other researchers outside of Outcome. The access to trial IPD will be limited to the researchers within Overcome for future full-scale research. However, the researchers might reconsider at the end of the study if the results from the thematic analysis and/or statistical analysis would be outside of our predictions.

REFERENCES:
- [Background] Vangsness L, Voss NM, Maddox N, Devereaux V, Martin E. Self-Report Measures of Procrastination Exhibit Inconsistent Concurrent Validity, Predictive Validity, and Psychometric Properties. Front Psychol. 2022 Feb 24;13:784471. doi: 10.3389/fpsyg.2022.784471. eCollection 2022. PMID 35282217
- [Background] Pollak KI, Alexander SC, Tulsky JA, Lyna P, Coffman CJ, Dolor RJ, Gulbrandsen P, Ostbye T. Physician empathy and listening: associations with patient satisfaction and autonomy. J Am Board Fam Med. 2011 Nov-Dec;24(6):665-72. doi: 10.3122/jabfm.2011.06.110025. PMID 22086809
- [Background] Otermin-Cristeta S, Hautzinger M. Developing an intervention to overcome procrastination. J Prev Interv Community. 2018 Apr-Jun;46(2):171-183. doi: 10.1080/10852352.2016.1198169. PMID 29485388
- [Background] Mutter A, Kuchler AM, Idrees AR, Kahlke F, Terhorst Y, Baumeister H. StudiCare procrastination - Randomized controlled non-inferiority trial of a persuasive design-optimized internet- and mobile-based intervention with digital coach targeting procrastination in college students. BMC Psychol. 2023 Sep 12;11(1):273. doi: 10.1186/s40359-023-01312-1. PMID 37700387
- [Background] Johnson SU, Ulvenes PG, Oktedalen T, Hoffart A. Psychometric Properties of the General Anxiety Disorder 7-Item (GAD-7) Scale in a Heterogeneous Psychiatric Sample. Front Psychol. 2019 Aug 6;10:1713. doi: 10.3389/fpsyg.2019.01713. eCollection 2019. PMID 31447721
- [Background] Jochmann A, Gusy B, Lesener T, Wolter C. Procrastination, depression and anxiety symptoms in university students: a three-wave longitudinal study on the mediating role of perceived stress. BMC Psychol. 2024 May 16;12(1):276. doi: 10.1186/s40359-024-01761-2. PMID 38755730
- [Background] Harrer M, Cuijpers P, Schuurmans LKJ, Kaiser T, Buntrock C, van Straten A, Ebert D. Evaluation of randomized controlled trials: a primer and tutorial for mental health researchers. Trials. 2023 Aug 30;24(1):562. doi: 10.1186/s13063-023-07596-3. PMID 37649083
- [Background] Connolly SM, Vanchu-Orosco M, Warner J, Seidi PA, Edwards J, Boath E, Irgens AC. Mental health interventions by lay counsellors: a systematic review and meta-analysis. Bull World Health Organ. 2021 Aug 1;99(8):572-582. doi: 10.2471/BLT.20.269050. Epub 2021 Apr 29. PMID 34354312
- [Background] Beutel ME, Klein EM, Aufenanger S, Brahler E, Dreier M, Muller KW, Quiring O, Reinecke L, Schmutzer G, Stark B, Wolfling K. Procrastination, Distress and Life Satisfaction across the Age Range - A German Representative Community Study. PLoS One. 2016 Feb 12;11(2):e0148054. doi: 10.1371/journal.pone.0148054. eCollection 2016. PMID 26871572